CLINICAL TRIAL: NCT06694103
Title: The Effect of Reverse Kangaroo Care Position and ROP Position on Pain During Retinopathy Examination in Premature Infants
Brief Title: The Effect of Two Non-Pharmacological Methods on Pain During Retinopathy Examination
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinem Basdemir (Other)
Responsible Party: Sponsor-Investigator, Sinem Basdemir, Research Assistant, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EU-HEM-SB-01
Record Dates: First submitted 2024-11-09; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Retinopathy of Prematurity (ROP)
Keywords: Premature; Retinopathy Screening; Retinopathy of Prematurity (ROP); Reverse Kangaroo Care Position; Pain
MeSH Terms: conditions — Retinopathy of Prematurity; Premature Birth; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reverse Kangaroo Care Position Group (Experimental): The advantages of kangaroo care will be utilised in the ROP examination. By reversing the position of the baby's face to the mother's breast, a change in the traditional kangaroo care posture will be applied, called the reverse kangaroo care position. Premature infants will be placed on the examination table for ROP examination and the infants' clothes other than diapers will be removed. Mothers will lie on the examination table by removing their upper clothes and their infants will be positioned in the inverted kangaroo care position, with the infant's back resting between the mother's bare chest. The privacy of the mother and the infant will be ensured and the infant will be able to smell the mother's scent with a piece of clothing taken off by the mother.
  Interventions: Other: Reverse Kangaroo Care Position
- ROP Position Group (Experimental): The position is given while the premature infant is in the supine position with the presence of two people (mother and nurse). It is performed in two stages by positioning the lower and upper extremities of the premature infant. The feet and legs are in the lower extremities, and the arms and head are in the upper extremities. During the examination, the premature infant's head is in slight hyperextension so that the retinal maneuvers applied by the ophthalmologist can be easily performed. The nurse places the infant's own palms on the temporal region and supports the head by holding it with her hands, while the mother supports the infant by bringing the infant's legs together and pushing it towards her abdomen.
  Interventions: Other: ROP Position

INTERVENTIONS:
Other: Reverse Kangaroo Care Position — * Babies will be taken to the examination table and their clothes other than diapers will be removed.
  * Mothers will take off their upper clothes and lie on the examination table and position their babies in the reverse kangaroo care position, with the baby's back against the mother's bare chest.
  * Babies will be monitored with disposable probes from their right feet.
  * Video recording will be started. -While the position applied to the babies is maintained, the speculum will be placed in the eye by the ophthalmologist and the examination will be recorded on video from the beginning to end.
  * After the completion of both eye examinations, the position of the babies whose monitoring continues will be maintained while the video recording will be taken for another 1 minute. The SPO2, HR, PIPP-R score at the end of the 15th second before the examination, the first minute during the examination and the 30th second after the examination will be evaluated.
  Arms: Reverse Kangaroo Care Position Group
Other: ROP Position — * Babies will be taken to the examination table and monitored with disposable probes from their right feet.
  * The nurse will place the infant's own palms on the temporal region and hold them with her hands to support their head, while the mother will also support the infant by holding their legs.
  * The video recording will be started.
  * SPO2, HR, PIPP-R values will be recorded on video for one minute.
  * While the ROP position applied to the babies is maintained, the speculum is placed in the eye by the ophthalmologist and the examination begins.
  * SPO2, HR, PIPP-R evaluation at the 1st minute of the examination.
  * After the completion of both eye examinations, the babies whose monitoring continues will be kept in their positions and a video recording will be taken for another 1 minute.
  * The SPO2, HR values and PIPP-R pain score at the end of the 30 seconds after the examination will be evaluated.
  Arms: ROP Position Group

SUMMARY:
The goal of this randomized controlled trial is to determine the effect of reverse kangaroo care position and ROP (Retinopathy of Prematurity) position applied during ROP examination in premature infants on pain. The main questions it aims to answer are as follows:

1. Is the reverse kangaroo care position effective in reducing the pain of premature infants during the ROP examination?
2. Is the reverse kangaroo care position more effective in reducing the pain of premature infants compared to the ROP position during the ROP examination?

Researchers will determine the effect of reverse kangaroo care position and ROP position applied during premature retinopathy examination in premature infants with a gestational age of less than 34 weeks on pain in infants.

* The infants of parents who volunteer to participate in the study will be divided into two groups as Reverse Kangaroo Care Position group and ROP Position group according to randomization.
* From the infants whose pupils are sufficiently mydriasis and are taken to the examination table, premature infants in the ROP Position group will be given ROP position together with the nurse and the parent.
* Premature infants in the Reverse Kangaroo Care Position group will be given reverse kangaroo care position.
* Video recording will be made during the given positions.
* The effects of the applied positions on pain will be determined as a result of the measured parameters before, during and after the examination.

DETAILED DESCRIPTION:
* 84 premature infants that meet the sample criteria will be determined.
* Randomization will be performed and premature babies will be assigned to the Reverse Kangaroo Care Position (Group 1) and Rope Position (Group 2) groups.
* The purpose of the study will be explained to the mother by meeting her and written consent will be obtained.
* The Premature Identification Form, which includes information about the infant, will be filled out.

According to the groups to which the premature infants who were randomized were assigned;

One minute before the examination;

1. The infants will be placed on the examination table and one drop of %0.5 alcaine (proparacaine HCl) topical anesthetic eye drops will be applied to both eyes of the premature infantss assigned to both groups by the neonatal intensive care nurse.
2. The pulse oximetry probe will be attached to the infants' right feet and monitored.
3. The infants will be positioned according to the group they are assigned to.
4. Video recording will be started one minute before the examination and will continue until 1 minute after the examination.
5. In order to evaluate the SPO2, KTA, PIPP-R values of all groups at the 15th second before the examination, the infant will be recorded on video for one minute.

During the Examination; In the Reverse Kangaroo Care Position Group;

1. While the reverse kangaroo care position applied to the infants is maintained, the speculum is placed on the eye by the ophthalmologist and the video recording will continue throughout the examination from the moment the examination begins
2. The SPO2, KTA, PIPP-R in the 1st minute of the examination will be recorded for evaluation

In the ROP Position Group;

1. While the ROP position applied to the babies is maintained, the speculum is placed on the eye by the ophthalmologist and the video recording will continue throughout the examination from the moment the examination begins
2. The SPO2, KTA, PIPP-R in the 1st minute of the examination will be recorded for evaluation

At the end of the examination;

1. After the completion of both eye examinations, the video recording will continue for 1 more minute while the positions of the babies whose monitoring continues are maintained
2. The video recording will end 1 minute after the examination ends
3. The infant's SPO2, KTA, values, PIPP-R pain score will be evaluated and recorded
4. . The aim is to record the infant's SPO2 and KTA values at 30 seconds so that the PIPP-R pain score can be evaluated later.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <34 weeks,
* Birth weight ≤ 2500 grams,
* No painful interventions at least 1 hour before the ROP examination,
* Fed at least 1 hour before the ROP examination,
* Premature infants whose parents consented to participate in the study.

Exclusion Criteria:

* Having a condition that prevents pain assessment (intracranial hemorrhage, neuromotor developmental delay etc.)
* Any congenital anomaly (eye, neurological, etc.),
* Have a diagnosed hearing problem,
* A different painful procedure was performed at least one hour before the ROP examination,
* Administration of an analgesic/sedative medication before the examination,
* Premature infants whose parents did not consent to participate in the study.

Ages: 28 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Premature Introductory Information Form: | Pre-intervention
  It was prepared by the researcher to determine the characteristics of the premature babies participating in the study. It consists of seven questions including the baby's gender, gestational week, birth weight, postnatal week, delivery method, birth head circumference and height measurement.
Premature Infant Follow-up Form | 15th minute before the examination; 1st minute during the examination, 30 seconds after the examination
  It consists of fields including the premature infant's heart rate, oxygen saturation values and PIPP-R score at the 15th second before the examination, the 1st minute during the examination and the 30 seconds after the examination.
Premature Infant Pain Profile Scale-Revised Form (PIPP-R) | 15th second before the examination; 1st minute during the examination, 30 seconds after the examination
  It is a Likert-type scale. In the scoring of the scale, items related to physiological and behavioral indicators are scored as 0, 1, 2 and 3 points for each variable. Items related to contextual indicators (behavioral status and gestational age) are scored as 3, 2, 1 and 0 points at the beginning of the pain assessment (before contact with the baby). According to PIPP-R, the infant's pain is evaluated based on the total score. In scoring the PIPP-R, behavioral and physiological indicators are scored at the end of the scale. Accordingly, if the infant receives a zero score (subtotal) from the general physiological and behavioral indicators, the contextual indicators are not scored. If the infant receives a score above zero from the initial parameters, the total score is obtained by including the contextual indicators in the scoring. The highest score of the PIPP-R is 21 for preterm infants and 18 for term infants (Stevens et al., 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Bal Yılmaz, Prof. Dr., Principal Investigator — Ege University
Locations (1):
- Izmır Provincial Health Directorate Bakircay University Cigli Regional Educational Hospital, Izmir, Menemen, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Only IPD used in the results publication. It will be shared later.